CLINICAL TRIAL: NCT04302350
Title: Nitrous Oxide for Identifying the Intersegmental Plane in Segmentectomy: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shijiang Liu, MD, doctor of The department of anaesthesiology and perioperate, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2019-SR-449
Record Dates: First submitted 2020-03-02; First posted 2020-03-10 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple; Lung Cancer
Keywords: pulmonary nodule; lung cancer; nitrous oxide; thoracoscopic anatomic segmentectomy
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Lung Neoplasms | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group75 (Experimental): According to preoperative 3D-CTBA evaluation of bronchial and vascular structure of pulmonary nodules and pulmonary segments, the target segmental bronchus, arteries and intra-segment veins were accurately identified and dissected by ligation or stapler cutting. After that, the anesthesiologist began to make preparations for the lung inflation. The portable nitrous oxide concentration detector (TD600-SH-B-N2O) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group75 set to N2O:O2=6:2). When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. This procedure took approximately 1 min, and then FiO2=1.0 was performed after the initiation of the OLV.
  Interventions: Procedure: nitrous oxide
- Group50 (Experimental): According to preoperative 3D-CTBA evaluation of bronchial and vascular structure of pulmonary nodules and pulmonary segments, the target segmental bronchus, arteries and intra-segment veins were accurately identified and dissected by ligation or stapler cutting. After that, the anesthesiologist began to make preparations for the lung inflation. The portable nitrous oxide concentration detector (TD600-SH-B-N2O) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group50 set to N2O:O2=4:4). When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. This procedure took approximately 1 min, and then FiO2=1.0 was performed after the initiation of the OLV.
  Interventions: Procedure: nitrous oxide
- Group0 (Active Comparator): According to preoperative 3D-CTBA evaluation of bronchial and vascular structure of pulmonary nodules and pulmonary segments, the target segmental bronchus, arteries and intra-segment veins were accurately identified and dissected by ligation or stapler cutting. After that, the anesthesiologist began to make preparations for the lung inflation. The portable nitrous oxide concentration detector (TD600-SH-B-N2O) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group0 set to O2=8). When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. This procedure took approximately 1 min, and then FiO2=1.0 was performed after the initiation of the OLV.
  Interventions: Procedure: nitrous oxide

INTERVENTIONS:
Procedure: nitrous oxide — During one-lung ventilation with an open chest, the nonventilated lung collapses initially due to elastic recoil, which quickly brings the lung down to its closing capacity. Remaining gas in the lung is then removed by absorption into the pulmonary capillary blood. The rapid diffusion properties of N2O（Blood gas distribution coefficient is 0.47）would be expected to speed lung collapse and so facilitate surgery. The previous study suggested that increasing the concentration of N2O in mixtures of N2O/O2 will lead to a faster rate of collapse. When using nitrous oxide in oxygen during lung ventilation, ongoing oxygen uptake by blood shunting will serve to increase the partial pressure of nitrous oxide in parts of the lung that are still expanded. This will soon result in a partial pressure gradient for nitrous oxide uptake also, with a consequent faster rate of lung collapse than would occur in a patient being ventilated with 100% oxygen.
  Other Names: oxygen

SUMMARY:
Lung cancer is currently one of the most common malignant tumors in the world. In recent years, with the popularity of high-resolution CT, more and more early-stage lung cancers have been found. Anatomic pneumonectomy is gradually popular because it can completely remove lung nodules and preserve lung function to the greatest extent. During the surgery, the precise and rapid determination of intersegmental border is one of the key technologies. Improved inflation-deflation method is currently the most widely used method in clinical practice. Previous studies demonstrated that increasing the concentration of nitrous oxide in mixtures of N2O/O2 will lead to a faster rate of collapse. The rapid diffusion properties of N2O would be expected to speed lung collapse and so facilitate surgery. This study was designed to explore three types of inspired gas mixture used during two-lung anesthesia had an effect on the intersegmental border appearance time during pneumonectomy and its feasibility and safety: 75% N2O (O2: N2O = 1: 3), 50% N2O (O2: N2O = 1: 1), 100% oxygen.

DETAILED DESCRIPTION:
This randomized parallel group trial enrolled lung cancer patients scheduled to receive thoracoscopic anatomic segmentectomy at The First Affiliated Hospital of Nanjing Medical University. When anesthesia induction was completed, intubation was carried out using an appropriate-size double-lumen endobronchial tube (DLT) and the position of the DLT was confirmed with fiberoptic bronchoscopy and adjusted as needed. OLV of the dependent lung with FiO2=1.0 was begun in the lateral position, by clamping the DLT to the nonventilated lung proximally and opening the distal port of the DLT lumen to the atmosphere. Tidal volumes were 5 mL/kg ideal bodyweight (male: height -100, and female: height - 105) without positive end expiratory pressure (PEEP). In order to avoid possible confounding effects of inhalation of volatile anesthetics on oxygenation, all subjects received total intravenous anesthesia.

According to preoperative 3D-CTBA evaluation of bronchial and vascular structure of pulmonary nodules and pulmonary segments, the target segmental bronchus, arteries and intra-segment veins were accurately identi-fied and dissected by ligation or stapler cutting. After that, the anesthesiologist began to make preparations for the lung inflation. The portable nitrous oxide concentration detector (TD600-SH-B-N2O) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group75 set to N2O:O2=6:2, Group50 set to N2O:O2=4:4, Group0 set to O2=8), avoiding the interference of the total gas flow. When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. This procedure took approximately 1 min, and then FiO2=1.0 was performed after the initiation of the OLV.

ELIGIBILITY:
Inclusion Criteria:

1、20 to 70 years of age; 2、early stage lung cancer（diameter of tumor consolidation ≤ 2cm, none evidence of lymph node or distant metas-tasis, c-stage ⅠA1 or ⅠA2）（active limited resection）； 3、 patients at high risk due to poor general condition who cannot undergo lobectomy (c-stage IA1 to IA3) (passive limited resection)

Exclusion Criteria:

1. a history of severe asthma or pneumothorax；
2. pulmonary bullae on chest CT；
3. patient refusal

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: cunming liu, Master, Study Chair — The First Affiliated Hospital with Nanjing Medical University; quan zhu, Doctorate, Study Director — The First Affiliated Hospital with Nanjing Medical University; shijiang liu, Attending physician, Study Director — The First Affiliated Hospital with Nanjing Medical University; wenjing yang, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; zicheng liu, Doctorate, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Wei Wen, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Jun Wang, Master, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three patients were excluded (1 refused to participate in the trial and 2 did not meet the inclusion criteria).
Groups:
- Group75: The target segmental bronchus, arteries and intra-segment veins were accurately identi-fied and dissected by ligation or stapler cutting. The portable nitrous oxide concentration detector (TD600-SH-B-N2O, tiandi shouhe, Beijing, Chi-na) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group75 set to N2O:O2=6:2). When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. FiO2=1.0 was performed after the initiation of the OLV.
  nitrous oxide: The rapid diffusion properties of N2O（Blood gas distribution coefficient is 0.47）would be expected to speed lung collapse and so facilitate surgery. The previous study suggested that increasing the concentration of N2O in mixtures of N2O/O2 will lead to a faster rate of collapse. When using nitrous oxide in oxygen during lung ventilation, ongoing oxygen uptake by blood shunting will serve to increase the partial pressure of nitrous oxide in parts of the lung that are still expanded. This will soon result in a partial pressure gradient for nitrous oxide uptake also, with a consequent faster rate of lung collapse than would occur in a patient being ventilated with 100% oxygen.
- Group50: The target segmental bronchus, arteries and intra-segment veins were accurately identi-fied and dissected by ligation or stapler cutting. The portable nitrous oxide concentration detector (TD600-SH-B-N2O, tiandi shouhe, Beijing, Chi-na) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group50 set to N2O:O2=4:4). When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. FiO2=1.0 was performed after the initiation of the OLV.
  nitrous oxide: The rapid diffusion properties of N2O（Blood gas distribution coefficient is 0.47）would be expected to speed lung collapse and so facilitate surgery. The previous study suggested that increasing the concentration of N2O in mixtures of N2O/O2 will lead to a faster rate of collapse. When using nitrous oxide in oxygen during lung ventilation, ongoing oxygen uptake by blood shunting will serve to increase the partial pressure of nitrous oxide in parts of the lung that are still expanded. This will soon result in a partial pressure gradient for nitrous oxide uptake also, with a consequent faster rate of lung collapse than would occur in a patient being ventilated with 100% oxygen.
- Group0: The target segmental bronchus, arteries and intra-segment veins were accurately identi-fied and dissected by ligation or stapler cutting. The portable nitrous oxide concentration detector (TD600-SH-B-N2O, tiandi shouhe, Beijing, Chi-na) was installed to detect N2O concentration (vol%), and then adjusted the anesthesia machine to the manual control mode. The flow of the selected gas mixture was set to 8L/min (Group0 set to O2=8). When the N2O concentration detector reached the predetermined gas concentration, and then the collapsed lung was re-expanded completely with controlled airway pressure under 20 cmH2O (1cm H2O=0.098 kPa) by the anesthesiologist. FiO2=1.0 was performed after the initiation of the OLV.
  nitrous oxide: The rapid diffusion properties of N2O（Blood gas distribution coefficient is 0.47）would be expected to speed lung collapse and so facilitate surgery. The previous study suggested that increasing the concentration of N2O in mixtures of N2O/O2 will lead to a faster rate of collapse. When using nitrous oxide in oxygen during lung ventilation, ongoing oxygen uptake by blood shunting will serve to increase the partial pressure of nitrous oxide in parts of the lung that are still expanded. This will soon result in a partial pressure gradient for nitrous oxide uptake also, with a consequent faster rate of lung collapse than would occur in a patient being ventilated with 100% oxygen.
Period: Overall Study
Arm/Group | Group75 | Group50 | Group0
Started | 26 | 26 | 26
Completed | 24 | 23 | 18
Not Completed | 2 | 3 | 8
Not completed — Physician Decision | 1 | 1 | 2
Not completed — Lack of Efficacy | 1 | 1 | 4
Not completed — Adverse Event | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group75 | Group50 | Group0 | Total
Number analyzed (Participants) | 24 | 23 | 18 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.04 (9.56) | 52.52 (10.86) | 50.50 (13.24) | 52.35 (11.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 12 | 46
  Male | 9 | 4 | 6 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  China | 24 | 23 | 18 | 65
body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.95 (3.04) | 21.61 (3.30) | 22.33 (2.38) | 22.29 (2.90)

OUTCOME MEASURES:

1. Primary Outcome: The Intersegmental Border Appearance Time During the Surgery
Description: The starting point of intraoperative expansion and collapse observation is the time when the lung tissue is completely expanded after blocking the relevant structure of the target segment; the end point is when a clear demarcation is formed between the target segment and the immediately-reserved lung segment, and this boundary does not follow significant changes over time), and the time was recorded in seconds (S).
Time Frame: The time of appearance of the intersegmental plane that can be performed satisfactorily by surgeons
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Group75 | Group50 | Group0
Number analyzed (Participants) | 24 | 23 | 18
seconds | 320.20 (65.89) | 552.39 (88.96) | 968.33 (85.53)

2. Other Pre Specified Outcome: The Incidence of Postoperative Complications and the Length of Hospital Stay
Description: Recording duration of surgery, the incidence of postoperative complications (including air leak, chylothorax, atelectasis, pulmonary embolism, pulmonary infection), total thoracic drainage, duration of drainage and postoperative hospital stay.
Time Frame: 2 weeks after surgery.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: After the patients finished the operation two weeks later
Description: Had intraoperative SPO2<90% during the perioperative period
Arm/Group | Group75 | Group50 | Group0
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/18
Other Adverse Events (participants affected / at risk) | 0/24 | 1/23 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group75 (N=24) | Group50 (N=23) | Group0 (N=18)
intraoperative SPO2<90% (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04302350/Prot_SAP_000.pdf